CLINICAL TRIAL: NCT03991078
Title: Pilot Clinical Study to Evaluate the Effect of Vitamin D on the Size of Fibroids in Women With Vitamin D Deficiency
Brief Title: Effect of Vitamin D on the Size of Fibroids in Women With Vitamin D Deficiency
Status: Completed | Type: Observational
Sponsor: Fundación IVI (Other)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: IIS-COL-2018-01; 1812-FIVI-100-AP (Registry Identifier: UAGI)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Size of the Uterine Fibroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitamin D supplementation in patients with uterine fibroids who present hypovitaminosis D to re-establish their normal serum values could stabilize the size of the uterine fibroids and thus prevent their growth or reduce their size thanks to the anti-proliferative action of Vitamin D on the myoma cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with at least one fibroid > 3 cm
* With hypovitaminosis D (25(OH)D < 30 ng/ml)
* BMI < 30
* No hormonal treatment in the 3 months prior to the ultrasound study

Exclusion Criteria:

* Black race
* Symptomatic fibroids subsidiary to hormonal or surgical treatment
* Desire of gestation in the next 6 months
* Presence of degenerating adenomyosis or fibroids
* Treatment with sexual hormones: mifepristone, aGnRH or any other medication that may interfere with fibroids.
* History of neoplasia of gynecological origin and/or existence of uterine malformations.
* Hypercalcemia or abnormal liver or kidney function is present

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with uterine fidroids and hypovitaminosis D
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
volume of the uterine fibroids | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, PhD, Principal Investigator — Fundación IVI
Locations (1):
- Fundacion IVI, Valencia, Spain

REFERENCES:
- [Derived] Orive A, Corachan A, Escrig J, Mascarell-Lopez MDM, Pellicer A, Monleon J, Ferrero H. Effect of low-dose vitamin D supplementation on uterine fibroid size in women with hypovitaminosis D: A nonrandomized pilot study. Int J Gynaecol Obstet. 2025 Nov;171(2):720-727. doi: 10.1002/ijgo.70271. Epub 2025 Jun 5. PMID 40470887